CLINICAL TRIAL: NCT00709787
Title: Epidemiological Study In Hypertensive Patients: Assessment Of Risk Factors Prevalence And Of Patients' Management
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A3841059
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Hypertension
Keywords: Epidemiology, hypertension, risk factors, coronary heart disease, patient management, compliance with medication
MeSH Terms: conditions — Hypertension; Coronary Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hypertensive Subjects undergoing primary prevention
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Usual Care — Normal care for hypertensive patients with risk factors for CHD

SUMMARY:
To assess the pattern of hypertension in the population in terms of presence of additional risk factors (ARF) and cardiovascular risk stratification.

DETAILED DESCRIPTION:
routine physician visits

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years old
* Patients with hypertension: newly diagnosed and /or already diagnosed and treated , whether at goal or not for the blood pressure level;
* Patients with no history of CHD/CVD

Exclusion Criteria:

* None

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Hypertensive Patients managed in primary care
Sampling Method: Non-Probability Sample
Enrollment: 899 (Actual)
Dates: Start 2008-06; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Description of hypertensive patients in terms of presence of associated cardiovascular (CV) risk factors (number of additional CV risk factors and frequency)

SECONDARY OUTCOMES:
Description of pattern of management of HT and CVD prevention, through lifestyle and use of drug therapies,
Estimate adherence to treatment using the Morisky Adherence Scale (MAS)
Estimation of hypertensive patients CV risk stratification based on ESH/ESC Hypertension Guidelines 2007 and to compare it with physicians' estimation of CV risk.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Pfizer Investigational Site, Varaždin, Croatia
- Pfizer Investigational Site, Prague, Czechia